CLINICAL TRIAL: NCT01125865
Title: Uncovered Self-expandable Metal Stent Versus DoubleLayer Plastic Stent for Malignant Hilar Stricture: a Prospective Randomized Multicenter Trial
Brief Title: Uncovered Self-expandable Metal Stent Versus Double Layer Plastic Stent for Malignant Hilar Stricture
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Tae Hoon Lee, Soon Chun Hyang University Cheonan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCH-2010-04
Record Dates: First submitted 2010-05-14; First posted 2010-05-19 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2010-05

CONDITIONS: Bile Duct Obstruction; Klatskin's Tumor
Keywords: Malignant hilar stricture
MeSH Terms: conditions — Cholestasis; Klatskin Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SEMS (Active Comparator): Self-expandable metallic stent will be inserted for the malignant hilar obstruction.
  Interventions: Device: SEMS insertion
- DLS (Active Comparator): DoubleLayer plastic stent (Olympus) will be inserted for malignant hilar obstruction.
  Interventions: Device: DLS insertion

INTERVENTIONS:
Device: SEMS insertion — Self-expandable metallic stent will be inserted for malignant hilar obstruction.
  Other Names: Bona stent; TaeWoong stent
  Arms: SEMS
Device: DLS insertion — DoubleLayer plastic stent will be inserted for malignant hilar obstruction.
  Other Names: Olympus DoubleLayer stent
  Arms: DLS

SUMMARY:
The overall median survival of nonresectable malignant hilar obstruction in most series has been less than 6 months. Most patients with malignant hilar obstruction present with advanced disease, making palliative endoscopic drainage the principal therapeutic option. However, the optimal endoscopic management strategy is contentious. Almost all of the published data comparing plastic and metallic stents relate to distal tumors (those of the pancreas, common bile duct and ampulla). Stent patency, complication rates, and cost-effectiveness have favored metallic stents when compared with plastic stents in patients with distal malignant obstruction expected to live at least 3 to 6 months.

There are few comparative study as to whether self-expanding metallic or plastic stent, especially DLS (double layer plastic stent) are preferable in the technical success, stent patency, and cost-effectiveness for palliating malignant hilar obstruction.

The study was designed to compare the the technical success, stent patency, and cost-effectiveness of self-expandable metal stent and DLS in patients with malignant hilar obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with malignant hilar obstruction

Exclusion Criteria:

* No written informed consent
* Patient with uncorrectable severe coagulopathy
* Indication for surgical operation
* Karnofsky score < 60%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Stent patency | Up to 2 years
  Interval time (d) from stent insertion to occlusion

SECONDARY OUTCOMES:
All cause complications | Up to 2 years
  Early or Late complications
  * asymptomatic hyperamylasemia
  * pancreatitis (mild/moderate/severe)
  * cholecystitis
  * cholangitis
  * recurrent jaundice
  * Internal migration
  * external migration
  * occlusion
Cost-effectiveness | Up to 2 years
  Total Cost for SEMS and DLS group
  * ERCP cost
  * Total ERBD cost (DLS or metal)
  * Total hospitalization cost
  * Cost for session x No. of session
  * Total (DLS vs. metal)cost /session
Mortality | Up to 2 years
Technical success | within 24 hr after stent insertion
  * Successful insertion of bilateral or unilateral stent insertion.
  * Time to adequate expansion (70% of maximal expanded diameter was dilated state) in metal stent ≤ 24 hrs
  * No stent migration within 24 hrs

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan, 23-20 Bongmyung-dong
  - Inje University Pusan Paik Hospital, Pusan, Busanjin-gu, Gaegeum-dong
  - Asan Medical Center, Seoul, Pungnap-2dong, Songpagu
  - Eulji University Hospital, Daejeon, Seo-gu, Dunsan-dong

REFERENCES:
- [Background] Tringali A, Mutignani M, Perri V, Zuccala G, Cipolletta L, Bianco MA, Rotondano G, Philipper M, Schumacher B, Neuhaus H, Schmit A, Deviere J, Costamagna G. A prospective, randomized multicenter trial comparing DoubleLayer and polyethylene stents for malignant distal common bile duct strictures. Endoscopy. 2003 Dec;35(12):992-7. doi: 10.1055/s-2003-44601. PMID 14648409
- [Background] Wagner HJ, Knyrim K, Vakil N, Klose KJ. Plastic endoprostheses versus metal stents in the palliative treatment of malignant hilar biliary obstruction. A prospective and randomized trial. Endoscopy. 1993 Mar;25(3):213-8. doi: 10.1055/s-2007-1010295. PMID 7686100
- [Background] de Groen PC, Gores GJ, LaRusso NF, Gunderson LL, Nagorney DM. Biliary tract cancers. N Engl J Med. 1999 Oct 28;341(18):1368-78. doi: 10.1056/NEJM199910283411807. No abstract available. PMID 10536130
- [Background] Yeoh KG, Zimmerman MJ, Cunningham JT, Cotton PB. Comparative costs of metal versus plastic biliary stent strategies for malignant obstructive jaundice by decision analysis. Gastrointest Endosc. 1999 Apr;49(4 Pt 1):466-71. doi: 10.1016/s0016-5107(99)70044-1. PMID 10202060
- [Background] Chang WH, Kortan P, Haber GB. Outcome in patients with bifurcation tumors who undergo unilateral versus bilateral hepatic duct drainage. Gastrointest Endosc. 1998 May;47(5):354-62. doi: 10.1016/s0016-5107(98)70218-4. PMID 9609426
- [Background] Davids PH, Groen AK, Rauws EA, Tytgat GN, Huibregtse K. Randomised trial of self-expanding metal stents versus polyethylene stents for distal malignant biliary obstruction. Lancet. 1992 Dec 19-26;340(8834-8835):1488-92. doi: 10.1016/0140-6736(92)92752-2. PMID 1281903
- [Background] Prat F, Chapat O, Ducot B, Ponchon T, Pelletier G, Fritsch J, Choury AD, Buffet C. A randomized trial of endoscopic drainage methods for inoperable malignant strictures of the common bile duct. Gastrointest Endosc. 1998 Jan;47(1):1-7. doi: 10.1016/s0016-5107(98)70291-3. PMID 9468416
- [Background] Cheng JL, Bruno MJ, Bergman JJ, Rauws EA, Tytgat GN, Huibregtse K. Endoscopic palliation of patients with biliary obstruction caused by nonresectable hilar cholangiocarcinoma: efficacy of self-expandable metallic Wallstents. Gastrointest Endosc. 2002 Jul;56(1):33-9. doi: 10.1067/mge.2002.125364. PMID 12085032